CLINICAL TRIAL: NCT05430971
Title: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) International Registry
Status: Recruiting | Type: Observational
Sponsor: Immune Oncology Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IMMONC0002
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN)
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | US Export: No

SUMMARY:
Blastic Plasmacytoid Dendritic Cell Neoplasm (BPDCN) is a very rare hematologic malignancy. Despite recent advances, at present there is no consensus on the optimal treatment of BPDCN. The optimal therapy of disease remains to be determined, and due to the rarity of cases, there is a need for international collaboration to collect data on BPDCN clinical presentations, diagnostics, treatment regimens and outcomes. Therefore, the objectives of this study are: (1) to build a large database of patients with BPDCN, (2) to investigate the characteristics and outcome of the disease with different treatment regimens, (3) to evaluate prognostic factors, and (4) to generate data-based prospective treatment recommendations.

DETAILED DESCRIPTION:
Blastic plasmacytoid dendritic cell neoplasm (BPDCN) is a rare hematologic malignancy. In 2008, it was recognized by the WHO as a distinct entity and separately listed in the group of acute myeloid leukemias and related precursor neoplasms.

The final diagnosis of BPDCN relies on a compatible immunophenotype. The triple positive CD4+CD56+CD123+ phenotype associated with negativity for lineage-specific markers is a minimum requirement for defining BPDCN. The highly specific marker BDCA2/CD303, as well as other plasmacytoid dendritic cell-associated antigens (e.g. TCL1 and CD2AP), might be of great support to exclude potential mimickers of BPDCN (acute myeloid and monocytic leukemias, precursor lymphoblastic T-cell leukemia/lymphomas and T- and NK/T cell lymphomas.

At present, there is no consensus on the optimal treatment of BPDCN. The majority of patients receive multi-agent chemotherapy with AML or ALL treatment regimens, while a few patients undergo allogeneic haematopoietic stem cell transplantation (HSCT). In recent years, different novel and innovative therapies are in development to target surface molecules in BPDCN. The patients are still in need of better treatments and the optimal therapy of disease remains to be determined.

This is a multicenter, international prospective and retrospective registry with the aim of collecting data of patients with a diagnosis of BPDCN globally.

Patients will be recruited directly by the national study groups / participating centers.

Participating centers will collect and verify informed consent of all prospective patients enrolled at their center.

The following data will be collected through questionnaires:

1. Patient characteristics
2. BPDCN characteristics
3. Treatment details
4. Outcomes
5. Cause of death
6. End of data collection

Quality control and data management will be conducted by the Immune Oncology Research Institute.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of BPDCN
* Signed informed consent form for prospective patients

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with BPDCN diagnosed since 01.01.2010
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2032-07 (Estimated); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Time from diagnosis to death

SECONDARY OUTCOMES:
Complete remission rate | 5 years
  The proportion of patients with complete remission
Mean duration of the first remission | 5 years
  Time from first remission to disease progression or death
Event-free survival | 5 years
  Time from diagnosis to occurrence of a complication

CONTACTS AND LOCATIONS:
Overall Officials: Astghik Voskanyan, MD, Principal Investigator — Immune Oncology Research Institute, Yerevan, Armenia; Gevorg Tamamyan, MD, PhD, DSc, Study Director — Immune Oncology Research Institute, Yerevan, Armenia
Locations (20):
- United States (3):
  - Sylvester Comprehensive Cancer Center, University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Seattle Children's Cancer and Blood Disorders Center, Seattle, Washington
- Hematology Center named after prof. R. Yeolyan, Yerevan, Yerevan, Armenia
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - Children's Hospital of Eastern Ontario, University of Ottawa, Ottawa, Ontario
- Cyprus Society of Haematology, Nicosia, Cyprus
- Oncology Center, Mansoura University Faculty of Medicine, Al Mansurah, Egypt
- M. Iashvili Children's Central Hospital, Tbilisi, Georgia
- Department of Medical Oncology, Dr. B.R.A Institute Rotary Cancer Hospital, All India Institute of Medical Sciences, New Delhi, India
- Pediatric Hematology Oncology, Children's Welfare Teaching Hospital, Medical City, College of Medicine, University of Baghdad, Baghdad, Iraq
- Italy (2):
  - University of Perugia - Azienda Ospedaliera Perugia, Perugia
  - Department of Biomedicine and Prevention, University of Rome Tor Vergata, Roma
- Department of hematology, Kuwait Cancer Control Center, Kuwait City, Kuwait
- Fundeni Clinical Institute, Department of Acute Leukemia, Bucharest, Romania
- China Medical University Children's Hospital, Taichung, Taiwan
- Turkey (Türkiye) (3):
  - Turkish Pediatric Cancer Registry, Ankara
  - Istanbul University, Oncology Institute, Istanbul
  - University of Health Sciences, Umraniye Research and Education Hospital, Pediatric Hematology and Oncology Department, Pediatric Bone Marrow Transplantation Unit, Istanbul
- Broomfield Hospital, Haematology Mid and South Essex University Hospitals Group, Chelmsford, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided